CLINICAL TRIAL: NCT02778412
Title: Determination of the Utility of Plasma Circulating Tumor DNA (ctDNA) Measurements for Detection of Thyroid Cancer in Patients Undergoing Diagnostic Fine Needle Aspirations of the Thyroid
Brief Title: ctDNA in Patients With Thyroid Nodules
Status: Terminated | Type: Observational
Why Stopped: Preliminary results indicated that this test had a number of false-negative results.
Sponsor: Pathway Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: Pathway Genomics-007
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Thyroid Cancer; Thyroid Nodules; Thyroid Adenoma; Thyroiditis
Keywords: Thyroid cancer; Thyroid nodules; Thyroid neoplasia; Thyroiditis
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Thyroiditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is drawn and DNA is purified from the plasma. The DNA is analyzed for circulating tumor DNA. The DNA will be stored for up to 10 years with the patient's permission.
Oversight: Data Monitoring Committee: No

SUMMARY:
When the DNA inside of human cells undergoes certain alterations (mutations), the cells may develop into a cancer. The cancer cells may shed this DNA into the blood stream. This circulating tumor DNA (ctDNA) can be detected by very sensitive, specialized laboratory tests. Measurement of ctDNA has been shown to be useful for following patients with known cancer. The purpose of this study is to examine blood specimens for the presence of ctDNA in individuals without known cancer who are scheduled to undergo a fine needle aspiration biopsy of the thyroid gland because of one or more thyroid nodules in order to see if the ctDNA test can detect a cancer at a very early stage. The results of this study should help define the role of ctDNA in the detection of early stage thyroid cancer and to define how sensitive it is (i.e. how well it picks up cancer when it is present) and how specific it is (i.e. how often is ctDNA found in patients with benign thyroid nodules).

DETAILED DESCRIPTION:
After the participants with thyroid nodules or other abnormalities have undergone the informed consent process, they will have 30 milliliters (approximately two tablespoons) of blood drawn. This will be done prior to the performance of the fine needle aspiration biopsy of the thyroid. If the patient has indicated a desire to receive the results of their test, they will receive a written description, as will their physician. The patients will be contacted yearly for up to 5 years by the study staff to learn whether they have been found to have a diagnosis of thyroid or other cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* presence of one or more thyroid nodules who are going to have a fine needle aspiration biopsy performed as part of their normal care.

Exclusion Criteria:

* Prior history of cancer excluding basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals 18 year of age or older without a prior diagnosis of cancer who are going to undergo a fine needle aspiration biopsy of the thyroid gland as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Utility of plasma ctDNA measurements to detect thyroid cancer | 1 year
  Correlation between plasma ctDNA results with pathology from the diagnostic fine needle aspiration biopsy of the thyroid gland.
Screening characteristics of ctDNA measurement in patients with and without thyroid cancer. | 1 year
  Determination of true positive, false positive and predictive values for using ctDNA measurements to detect thyroid cancer.

SECONDARY OUTCOMES:
Determination of incident rate of new thyroid or other cancers in patients who underwent initial measurement of ctDNA. | 5 years
  Subjects will be contacted yearly to obtain follow-up information regarding the development of thyroid or other cancer in order to see if the initial ctDNA measurement detected the cancer before it became clinically apparent.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D. Braunstein, M.D., Principal Investigator — Pathway Genomics; Anja Kammesheidt, PhD, Principal Investigator — Pathway Genomics
Locations (1):
- Thyroid & Endocrine Center of Florida, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The patient's physician will receive the results and the patients have the option to also receive the results.

REFERENCES:
- [Background] Pupilli C, Pinzani P, Salvianti F, Fibbi B, Rossi M, Petrone L, Perigli G, De Feo ML, Vezzosi V, Pazzagli M, Orlando C, Forti G. Circulating BRAFV600E in the diagnosis and follow-up of differentiated papillary thyroid carcinoma. J Clin Endocrinol Metab. 2013 Aug;98(8):3359-65. doi: 10.1210/jc.2013-1072. Epub 2013 Jun 20. PMID 23788690